CLINICAL TRIAL: NCT06760988
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy of CL22205 to Improve Menstrual Discomfort and Quality of Life
Brief Title: Efficacy of CL22205 to Improve Menstrual Discomfort and Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eetho Brands, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: EB/MH/CL22205/24
Record Dates: First submitted 2024-12-24; First posted 2025-01-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Menstrual Discomfort
Keywords: Quality of life

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CL22205 (Experimental): 200 mg - One capsule a day after breakfast for 135 days
  Interventions: Dietary Supplement: CL22205
- Placebo (Placebo Comparator): One Capsule a day after breakfast for 135 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: CL22205 — Experimental Dose: 200 mg, Mode: Oral, once daily after breakfast Duration: 135 days
  Arms: CL22205
Other: Placebo — Mode: Oral, once daily after breakfast Duration: 135 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of CL22205 to improve menstrual discomfort and quality of life in oligomenorrheic female subjects.

DETAILED DESCRIPTION:
A total of 80 oligomenorrheic female subjects aged between 25 and 35 years will be included in the study. Assessment of inclusion and exclusion criteria will be done based on clinical and laboratory investigations. The eligible subjects will be randomized as per the computer-generated randomization list. The subjects will be assigned to either CL22205 - 200 mg or placebo arm at 1:1 ratio. The subjects will be instructed to take one capsule a day after breakfast for 135 days. Apart from primary and secondary outcomes, the study will also record the vital signs and adverse events to evaluate the herbal composition's safety and tolerability. The safety assessment of the CL22205 will also include routine laboratory investigations on blood, urine and clinical chemistry at screening and the final visit of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Oligomenorrheic females (Menstrual cycle duration between 36-45 days), aged between 25 and 35 years and with a Body Mass Index (BMI) between 20 to 29.9 kg/m2.
* Subjects with maximum pain intensity ≥40 mm on a 100 mm VAS for at least 2 menstrual cycles before participating in the study.
* Subjects with normal thyroid profile.
* Subjects who are non-smokers and non-alcohol user.
* Subject understands the study procedures and provides signed informed consent to participate in the study.
* Females of childbearing potential who are sexually active must agree to use adequate non-hormonal contraception during the study.
* Normal vital signs, including electrocardiogram (ECG) and laboratory evaluations (including clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory or the results are deemed not clinically significant for inclusion into this study by the investigator.

Exclusion Criteria:

* History of any gynaecological disorders which effects the study indication.
* History of cerebrovascular disease, thrombo-embolic disorders, heart attack, or angina at any time or thrombophlebitis within the last 5 years, on anti-coagulant or anti-platelet drugs on a daily basis for any conditions.
* Subjects who had any hormonal therapy, metformin or any other herbal products in the past 3 months.
* Hypothyroidism, hyperthyroidism, hyperprolactinemia, Cushing's syndrome and congenital adrenal hyperplasia, following a special diet for the past 3 months, taking drugs affecting insulin sensitivity or lipid and hormonal profiles, including glucocorticoids, ovulation-stimulating drugs, anti-obesity, anti-diabetes, anti-hypertensive, anti-estrogenic, anti-androgenic during the last 3 months (except the usual drugs of the subjects).
* Active gall bladder disease, gynaecological or breast surgery in the last 6 months.
* Subjects underwent hysterectomy.
* History of breast, endometrial, other gynaecological cancer at any time or other cancer within the last 5 years.
* Pregnant and lactating mothers.
* History of hypersensitivity reactions attributed to investigational product (IP) or its components or related products.
* History of positive hepatitis, including Hepatitis B surface antigen or Hepatitis C virus (HCV) antibodies or subjects with human immunodeficiency virus (HIV) and /or syphilis.
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol.
* Participated in a clinical study with an investigational drug or biologic within the last 60 days.
* Any condition that in opinion of the investigator, does not justify the subjects' participation in the study.
* Subjects who are being treated for liver cancer or cirrhosis, chronic renal failure, congestive heart failure.
* Subjects with a systemic disease including tuberculosis, leucosis, collagenosis, multiple sclerosis or other autoimmune diseases.
* Subjects with a high blood pressure at screening (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg).
* Consumption of recreational drugs (such as cocaine, methamphetamine, marijuana, etc.) or psychiatric drug users.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Oligomenorrheic females (Menstrual cycle duration between 36-45 days)
Enrollment: 80 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2025-10-05 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to the end of the study period in: The Menstrual Symptoms Questionnaire (MSQ) scores | Day 1, Day 45 (±10 days), Day 90 (±10 days), Day 135 (±10 days)
  The Menstrual Symptom Questionnaire (MSQ) is a tool used to assess the severity and type of menstrual symptoms experienced by individuals. This questionnaire includes 24 items, where subjects will be instructed to indicate the degree to which they experience the symptom by selecting one of the five responses [Never (N), Rarely (R), Sometimes (S), Often (O). and Always (A).
  The first 24 items are characteristics of either spasmodic or congestive dysmenorrhea. The type of dysmenorrhea indicates the order of scoring for each item. Items designated as S (Spasmodic), score as indicated by numbers 1-5. Items designated as C (Congestive), reverse scoring.
  For the twenty-fifth item subjects will be instructed to read the descriptions of two types of menstrual discomfort and select the type that most closely fits their experience. The subjects with spasmodic dysmenorrhea will receive higher total scores while those with congestive dysmenorrhea will receive lower total scores.

SECONDARY OUTCOMES:
Change from baseline to the end of the study period in: Ovarian Follicular analysis | Day 1 & Day 135 (±10 days)
  using USG
Change from baseline to the end of the study period in: Serum levels of FSH and LH | Day 1 & Day 135 (±10 days)
  Biomarkers
Change from baseline to the end of the study period in: Scores of subjective self-assessment on hair quality | Day 1, Day 45 (±10 days), Day 90 (±10 days), Day 135 (±10 days)
  This is a subjective measurement of hair quality by considering the hair fall rate, assessed based on the number of hair strands shed per day, with scores ranging from 1 to 5 (score 1: >100strands, score 2: 50-100 strands, score 3: 30-50strands, score 4: 10-30 strands and Score 5: Less than 10 (indicating best possible condition).
  The hair texture assessment, ranges from 1 to 5 (score 1: Rough and frizzy (worst possible condition) to 5: Very soft (best possible condition.)) The hair volume ranges from 1 to 5, (Score 1: Very low volume (worst possible condition) to Score 5: Excellent volume (best possible condition.)) The hair fall grading ranges from 0 to 5, (Score 0: No itching (best possible condition); Score 5: Very severe itching.))
Change from baseline to the end of the study period in: Scores of Global Acne Grading system for acne | Day 1, Day 45 (±10 days), Day 90 (±10 days), Day 135 (±10 days)
  The Global Acne Grading System (GAGS) is a widely used method to assess the severity of acne vulgaris. This system grades the acne present on face, chest, and upper back by considering 7 locations viz; the forehead, right cheek, left cheek, nose, chin, and chest and upper back combined. Each acne lesion will be graded as no lesions (grade 0) a comedone (grade 1), papule (grade 2), pustule (grade 3), or nodule (grade 4).The local score for each anatomic area was determined by multiplying the grade of the most severe lesion with an area specific factor (1 to 3), and then summation of all 7 local scores represents the total acne severity score.
  Acne severity was graded as none (total score, 0 points), mild (total score, 1-18 points), moderate (total score, 19-30 points), severe (total score, 31-38 points), and very severe (total score >38 points).
Change from baseline to the end of the study period in: Menstrual distress questionnaire (MDQ) | Day 1, Day 45 (±10 days), Day 90 (±10 days), Day 135 (±10 days)
  The Menstrual Discomfort Questionnaire (MDQ) consists of 46 item self-reported inventory used to assess the premenstrual and menstrual symptoms measured at three time points: "Most Recent Flow" (menstrual phase), "Four Days Before" (premenstrual phase), and "Remainder of Cycle" (intermenstrual phase). For each item, respondents rate their experience using a 5-point scale: where 0 means, no experience of symptom, 1: Present, mild 2: Present, moderate 3: Present, strong 4: Present, severe. Respondents select the category that best describes their experience. The 46 items are grouped into 8 domains (Pain, Water Retention, Autonomic Reactions, Negative Affect, Impaired Concentration, Behavior Change, Arousal, and Control). Raw scores for each domain are calculated for the three phases and then converted to T-scores. Higher T-scores indicate greater distress.
Change from baseline to the end of the study period in: Regularity in menstrual cycles (duration between two menstrual bleedings) | Day 1, Day 45 (±10 days), Day 90 (±10 days), Day 135 (±10 days)
  menstural regularity
Change from baseline to the end of the study period in: Serum levels of AMH, total testosterone and Progesterone | Day 1 & Day 135 (±10 days)
  Biomarkers
Change from baseline to the end of the study period in: Serum levels of SHBG, 17β Estradiol (E2), and Prostaglandin F2 alpha (PGF2 alpha). | Day 1 & Day 135 (±10 days)
  Biomarkers
Change from baseline to the end of the study period in: Female Sexual Function Index (FSFI) | Day 1, Day 45 (±10 days), Day 90 (±10 days), Day 135 (±10 days)
  The FSFI was developed as a brief, easy-to-administer, self-report tool for assessing key dimensions or domains of sexual function and quality of life in various populations of women. Female Sexual Function Index (FSFI), a widely used tool with six domains (Arousal, Desire, Orgasm, Lubrication, Satisfaction, and Pain). The total FSFI score ranges from minimum score of 2 and maximum score of 36. Greater Scores indicates better sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Varuni B.G, Principal Investigator — Consultant

IPD SHARING:
Plan to Share IPD: No